CLINICAL TRIAL: NCT02854020
Title: Comparison of Inflight First Aid Performed by Cabin Crew Members and Medical Volunteers
Status: Completed | Type: Observational
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, JUNGHA KIM, Principal Investigator, Seoul National University
Other Study IDs: SeoulNU
Record Dates: First submitted 2016-07-18; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Emergency
Keywords: Aircraft; Emergency; First aid; Cabin crew; Burn; Cardiac arrest
MeSH Terms: conditions — Emergencies; Burns; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- An asian airline

SUMMARY:
Since the number of air travelers, including the elderly and passengers with an underlying disease, is increasing every year, the number of inflight emergency patients is expected to increase as well. The investigators attempted to identify the incidence and types of inflight medical emergencies and analyze the first aid performed by cabin crew members or medical volunteers in flights by an Asian airline. The investigators also investigated the causes of inflight deaths and aircraft diversions.

ELIGIBILITY:
Inclusion Criteria:

* Inflight medical emergencies from 2009 to 2013

Exclusion Criteria:

* Events that occurred before takeoff or after landing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inflight medical emergencies from 2009 to 2013
Sampling Method: Non-Probability Sample
Enrollment: 2818 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Types of inflight medical emergencies confirmed by reviewing cabin reports submitted by cabin crew and medical records submitted by medical volunteers | 5 years (events during inflight, excluding events that occured before takeoff or after landing)
  Types of inflight medical emergencies were created according to the initial symptoms of passengers (e.g. syncope, trauma)

SECONDARY OUTCOMES:
Incidence of inflight medical emergencies confirmed by reviewing cabin reports submitted by cabin crew and medical records submitted by medical volunteers | 5 years (events during inflight, excluding events that occured before takeoff or after landing)
  Incidence in inflight emergencies/million passengers
The causes of inflight deaths and aircraft diversions confirmed by reviewing cabin reports submitted by cabin crew and medical records submitted by medical volunteers | 5 years (events during inflight, excluding events that occured before takeoff or after landing)
  The causes of deaths and diversions were confirmed by types of inflight